CLINICAL TRIAL: NCT02769143
Title: Effects of Whole Body Vibration and Pilates Method on Bone Mineral Density in Postmenopausal Women: a Randomized, Controlled, Clinical Trial
Brief Title: Effects of Whole Body Vibration and Pilates on Bone Mineral Density in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Norte do Paraná (Other)
Responsible Party: Principal Investigator, Lais Campos de Oliveira, doctoral student in Sciences Program Rehabilitation, Universidade Norte do Paraná
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1.032.182
Record Dates: First submitted 2016-05-07; First posted 2016-05-11 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Bone Mineral Density Quantitative Trait Locus 3
Keywords: Postmenopausal; Bone Density; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Whole-Body Vibration Group (WBV) (Experimental): Will be exposed to five minutes on a vibrating platform (Oscillating Platform Semi-Professional Horizontal - Arktus, Cascavel, Brazil), this type of platform vibrates through an anteroposterior axis, causing the right and left sides alternate horizontally denominated: alternating side vibration platforms, will be performed three times per week on alternate days (5 minutes). a frequency of 20 Hz (1 = 1 Hz oscillation / second) and a magnitude of 3.2 g (1 g = 9,81 m / s gravity) is used. The volunteers will be guided to stand on the platform with semi-flexed knees, barefoot and apart about hip width.
  Interventions: Other: Whole-Body Vibration
- Pilates Group (PG) (Experimental): Will be exposed to 60 minutes, held three times a week on alternate days. Pilates equipment used for the exercises are: Combo Chair, Cadillac Trapeze, Ladder Barrel, Reformer Universal, Step Barrel and Wall Unit. Will be selected for this study, 21 strengthening exercises and stretching to the main body segments. All exercises are performed in a series of ten repetitions with one minute interval between exercises. To determine the level of effort and consequently to changing loads, will be used verbal command according to the Borg CR10 scale. The level of effort will be maintained during the session heavy (Borg between 5 and 6).
  Interventions: Other: Pilates
- Control Group (CG) (No Intervention): The control group will be instructed to maintain their usual activities both in relation to their daily activities, dietary habits, failure to use drugs that can influence the increase in bone mass and participate in monthly meetings to address on issues osteoporosis and postmenopausal women. After the end of the interventions with WBV and GP groups, GC volunteers will be invited to also perform whole body vibration for six months. Exposure of vibration will be for five minutes on a vibrating platform, three times per week on alternate days. a frequency of 20 Hz (1 = 1 Hz oscillation / second) and a magnitude of 3.2 g (1 g = 9,81 m / s gravity) is used. Likewise which was offered for the WBV group.

INTERVENTIONS:
Other: Whole-Body Vibration — Will be performed six months of WBV exercises
  Other Names: Whole-Body Vibration Exercise
  Arms: Whole-Body Vibration Group (WBV)
Other: Pilates — Will be performed six months of Pilates exercises
  Other Names: Pilates Exercise
  Arms: Pilates Group (PG)

SUMMARY:
Women in the postmenopausal period suffer hormonal changes that contribute to a number of negative factors to health, such as reduced bone mineral density and loss of muscle mass, which contribute to the increased incidence of falls and consequent risk of fractures. Among the possibilities to alleviate these symptoms are mainly drug treatment and the systematic practice of physical exercise. Exercise stands out for not offering adverse effects. One form of exercise that has been recently investigated is the whole body vibration, another form of exercise well accepted by the population is the Pilates method.

Taking into account the lack of literature on the benefits of vibration training; and also the Pilates method on bone mineral density, muscle strength, flexibility, postural balance, fear of falling and the quality of life of postmenopausal women, explains the importance of this work.

DETAILED DESCRIPTION:
Women in the postmenopausal period suffer hormonal changes that contribute to a number of negative factors to health, such as reduced bone mineral density and loss of muscle mass, which contribute to the increased incidence of falls and consequent risk of fractures. Among the possibilities to alleviate these symptoms are mainly drug treatment and the systematic and regular physical exercise. However, drug treatment primarily involves hormone replacement therapy, which is associated with increased risk of heart disease, stroke and breast cancer. Thus, exercise stands out for not offering adverse effects, however, when it comes to bone metabolism, it is not yet clear what type of exercise is the most effective for women in the postmenopausal period.

One form of physical exercise that has recently been investigated is the whole-body vibration (WBV), characterized by individual placement on a vibrating plate capable of transmitting vertical acceleration for the musculoskeletal system, however, the intensity (frequency and magnitude) ideal to allow increased bone metabolism has not been established and remain controversial.

Other forms of exercise have been recommended for postmenopausal women, such as those of muscular endurance. Exercises involving strength training, using weight can contribute to the improvement of bone mineral density of women in the postmenopausal period. Another form of exercise that also offers endurance is the Pilates method. However, the effects of this technique on bone mineral density, has not been investigated, despite having shown potential contribution on the variables pain, functional capacity and quality of life in postmenopausal women.

This study is justified because there are still shortages of literature and evidence about the benefits of vibration training; and also Pilates, on bone mineral density in postmenopausal women. There are also still little information about how much vibration training can influence muscle strength, flexibility, postural balance, fear of falling and the population's quality of life in question.

ELIGIBILITY:
Inclusion Criteria:

* Clinical confirmation of postmenopausal for at least 12 months
* Not exercise practitioner for at least six months
* Agreement not to do another type of exercise during the search
* Ability to perform activities of daily living without assistance
* Medical certificate stating fitness to practice physical exercise; cognitive state ≥19 according to the Mini-Mental State Examination (MMSE)

Exclusion Criteria:

* Musculoskeletal disorders in the spine or the lower limbs in the last six months; fracture in the spine or lower limbs after 40 years of age
* Prosthesis in the lower limbs or implants in the spine; Secondary causes of loss of bone mass
* Other metabolic bone diseases or diseases affecting bone metabolism; history of cancer in the last five years; vascular changes
* Epilepsy or seizures; arrhythmia; Pacemaker use; eye disease affecting the retina
* Cardiorespiratory diseases; diseases in the neuromuscular system; labyrinthitis or lightheadedness
* Hospitalization in the last six months for surgical reasons; alteration of Thyroid, drinking alcohol
* Smoking
* Use of supplements such as calcium or vitamin D, or containing isoflavones
* Medication to increase bone mineral density or increased muscle mass in the last 12 months
* Inability to tolerate 5-minute whole body vibration

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-05; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Bone mineral density | six months
  To analyze the bone mass of the femoral neck and lumbar spine (L1-L4) will use the device-ray Absorptiometry Dual Energy X (DXA) HOLOGIC, DQR-1000 PLUS model. The technique is based on the attenuation by the patient's body, a radiation beam generated by an X-ray source with two power levels, and exposure to radiation is lower than that of a conventional X-ray examination. The technique allows to estimate bone mass in whole and body segment. The results are transmitted to the computer that is connected to the device.
  Bone mineral density (BMD) is expressed as absolute values (g / cm2 grams of bone mineral content per area or analyzed bone cm2).

SECONDARY OUTCOMES:
Muscle strength | six months
  The muscle strength of the lower limbs will be measured through the movements of extension and knee flexion (concentric / concentric) with the Biodex System 4.0 equipment (Biodex Medical Systems, Shirley, NY), using to the extent the number less preferably with three tries, five repetitions each at an angular velocity of 60 and 180 degrees per second (60º / s and 180º / s). Among the attempts will be respected 30 seconds of rest. Will be considered for analysis, peak isokinetic torque (PT) and total work (TW), expressed in newtons per meter (Nm) and joules (J) respectively. Prior to the test, the device will be calibrated following the manufacturer's standards. The heating will be held for five minutes in an upright stationary bike with light load (25 watts) and comfortable speed (50 revolutions per minute).
Flexibility | six months
  For analysis of the flexibility instrument will be used Fleximeter (Institute Code Research, São Paulo, Brazil), for the flexion and extension of the trunk. For the trunk flexion movement, the volunteer should remain standing, with extended knees, bent arms, hands resting on the neck. Fleximeter will be positioned laterally in the thoracic region, with the display facing the evaluator, the right side of the trunk. With voluntary upright, the evaluator should reset the Fleximeter and later support the hands on the knees of voluntary in order to preclude the bending thereof. Following the voluntary hold the maximum flexion of the trunk, holding this position for a few seconds so that the evaluator performs the reading range of motion. For the trunk extension movement, the procedures will be the same, however, voluntary hold the maximum extension of the trunk.
Postural balance | six months
  For assessment of postural balance static will be used a force platform, BIOMEC 400 model (EMG System of Brazil Ltda., São Paulo). The assessor will explain the test procedures for voluntary, which will have a moment of familiarization with the equipment and the test will run. Following the participants carry out the balancing task with bipedal support, (with eyes open and eyes closed), semi-tandem (with eyes open and then with eyes closed) and one-leg (with eyes open). 30 seconds three attempts will be made with equal rest time (30 seconds) there between. The order of execution of each task (bipedal, single leg and semi-tandem) will be randomized. For further analysis of the data, the average of attempts is used. The volunteers should be barefoot, loose arms and relaxed beside the body and the following head positioned horizontally at ground level, being oriented to look at a fixed target (white paper circle with 3 cm in diameter) positioned in the wall at a distance of 2 meters
The Timed Up and Go test (TUG) | six months
  Will be used for analysis of functional mobility and the risk of falls. marking will be placed on the floor measuring three meters from the front of a chair with arms. The volunteer will be oriented that when said the word "already" should get up from the chair, normally walk to the end marker, turn and walk back to the chair, sitting down again. The timer will be triggered to be said the word "already" and stopped at the time the volunteer sit in the chair. The shorter the time taken for completion of this course, the better the result of the test (less than 10 seconds is considered low risk for falls; between 10 and 20 seconds, medium risk of falls; above 20 seconds a high risk of falls). Three attempts will be performed and only the best will be considered.
Fear Falls | six months
  The evaluation of the fear of falling will be held across the range Falls Efficacy Scale - International (FES-I) in your translated and adapted for the Brazilian population, consisting of 16 questions that identify concern about the possibility of falling in daily activities, outdoor activities and social participation, their total score ranges between 16 and 64 points, so that higher scores indicate greater concern about falling. It demonstrates good reliability and internal consistency with values similar to the original version, considered appropriate to assess the fear of falling in the population of elderly Brazilians.
Quality of life | six months
  For the quality of life will be used the Brazilian version of the SF-36 questionnaire. This questionnaire consists of 11 questions and 36 items covering eight components (domains or dimensions), represented by functional capacity (ten items), physical (four items), pain (two items), general health (five items), vitality (four items), social functioning (two items), emotional aspects (three items) and mental health (five items). The individual receives a score in each domain, ranging from 0 to 100, 0 being the worst score and 100 the best.

CONTACTS AND LOCATIONS:
Overall Officials: Deise A de Almeida Pires-Oliveira, Doctor, Principal Investigator — Universidade Norte do Paraná
Locations (1):
- Universidade Norte do Paraná, Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No